CLINICAL TRIAL: NCT01719575
Title: A Double-blind, Randomized, Two-way, Cross-over Study for Evaluating Motilitone on Gastric Motor Function in Healthy Volunteers
Brief Title: Clinical Trial of Motilitone on Gastric Motor Function in Healthy Volunteers
Acronym: DA-9701
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: DA9701_GA_IV
Record Dates: First submitted 2012-10-26; First posted 2012-11-01 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Female and Male

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motilitone (Other): take motilitone 30mg three times daily for the first week After 7 day wash-out period, take placebo three times daily for the second week
  Interventions: Drug: Motilitone
- Placebo (Other): take placebo three times daily for the first week After 7 day wash-out period, take motilitone 30mg three times daily for the second week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Motilitone
  Arms: Motilitone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects of Motilitone and placebo on gastric volumes, gastric emptying, small bowel transit and colon transit in female and male healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* no gastrointestinal symptoms
* no organic lesion such as gastrointestinal malignancies, erosive esophagitis, reflux esophagitis, erosive gastroduodenitis, gastric or duodenal ulceration after having normal upper abdominal endoscopy
* written informed consent

Exclusion Criteria:

* pregnant, breast-feeding female,those of childbearing age who were not using an approved method of contraception
* history of abdominal surgery that may influence gastrointestinal motility
* gastrointestinal hemorrhage, mechanical ileus, enterobrosis
* irritable bowel syndrome, inflammatory bowel disease
* severe disturbance of liver, kidney, heart,lung,blood and endocrine
* psychoneurosis, alcoholism, drug dependence
* medications that may alter evaluation of Motilitone including antibiotics,corticosteroids, NSAID within 1 month, prokinetics, H2 blocker, PPI, anticolines, erythromycin, antidepressive agents withing 2weeks

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
gastric fuction of Motilitone | 3 weeks
  gastric emptying time on day 4 by scintigraphic imaging
gastric function of Motilitone | 3 weeks
  fasting and postprandial gastric volume on day 7 by single photon emission computed tomography

SECONDARY OUTCOMES:
adverse events of Motilitone | 3 weeks
small bowel function of Motilitone | 3 weeks
  small bowel transit time on day 4 by scintigraphic transit measurement
Colon function of Motilitone | 3 weeks
  colon transit time on day 4 and 7 by KUB

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Gyu Choi, Ph.D., Principal Investigator — Seul St.Mary's hospital
Locations (1):
- the Catholic university of korea college of Medicine, Seoul St.Mary's hospital, Banpo-dong, Seocho-gu, Seoul, South Korea